CLINICAL TRIAL: NCT02619851
Title: A Phase II Clinical Trial to Evaluate the Safety and Efficacy of ALLO-ASC-DFU for Second Deep Degree Burn Injury Subjects: Controlled, Parallel, Multicenter
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of ALLO-ASC-DFU for Second Deep Degree Burn Injury Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-ASC-BI-201
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Burn Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALLO-ASC-DFU (Experimental): Allogeneic mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-DFU
- Conventional Therapy (Active Comparator): Typical therapy conducted for burn injury patients
  Interventions: Device: Conventional Therapy

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Dressing for Second Deep degree Burn injury
  Other Names: Allogeneic mesenchymal stem cells
  Arms: ALLO-ASC-DFU
Device: Conventional Therapy — Typical therapy conducted for burn injury patients
  Arms: Conventional Therapy

SUMMARY:
This clinical trial is a Phase II controlled, parallel, open-label trial, designed to test the efficacy and safety of ALLO-ASC-DFU and conventional therapy in Deep Second-degree burn wound subjects.

DETAILED DESCRIPTION:
ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating Deep Second-degree burn wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age and older.
2. Subjects who have deep second-degree burn wound ≥100cm^2.
3. TBSA(Total burn surface area) ≤ 30%
4. Negative for Urine beta-HCG for women of childbearing age.
5. Subject is able to give written informed consent prior to study start and comply with the study requirements.

Exclusion Criteria:

1. Subject who have been enrolled in another clinical study within 30 days of screening.
2. Subjects who are allergic or have a hypersensitive reaction to bovine-derived proteins or fibrin glue.
3. Subjects who are receiving steroids, immunosuppressive, or anticoagulant for long term
4. Subjects with active infection.
5. Subjects with hemorrhagic and hemocoagulative disease.
6. Subjects who are unwilling to use an "effective" method of contraception during the study.
7. Subjects who have a history of malignant tumor within the last five years, or is currently undergoing.
8. Subjects who are pregnant or breast-feeding.
9. Subjects who are considered to have a significant disease which can impact the wound healing by the investigator
10. Burn wound is present on any part of the face.
11. Subjects who are considered not suitable for the study by the investigator.
12. Subjects who are not able to understand the objective of this study or to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Time of re-epithelialization | Follow up to 12 weeks
  Time of re-epithelialization

SECONDARY OUTCOMES:
Safety (laboratory tests and adverse events) | Follow up to 12 weeks
  Clinically measured abnormality of laboratory tests and adverse events
Burn Scar Index | Follow up to 12 weeks
  Vancouver Burn Scar Scale
healing status of the wound evidenced by photography | follow up to 12 weeks
  healing status of the wound evidenced by photography

CONTACTS AND LOCATIONS:
Overall Officials: Wook Chun, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym university Medical Center, Seoul, South Korea